CLINICAL TRIAL: NCT05622006
Title: The Effects of Interrupting Sedentary Behaviour With Different Frequencies of Physical Activity on Cardiometabolic- and Cardiovascular Risk Factors
Brief Title: Effect of Interrupting Sedentary Time With Different Frequencies of Physical Activity on Cardiometabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Jostein Steene-Johannessen, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GENSED
Record Dates: First submitted 2022-11-04; First posted 2022-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sedentary; Cardiometabolic Syndrome; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will be conducted as randomized controlled crossover trials involving 4 different trial conditions in each of the studies. Randomization will be stratified based on sex. The order of trials will be assigned randomly by a third party using a computer software.
  After pre-testing and familiarization (visit 1), the participants will undergo 4 different trial conditions of 7 hours. The trials are all iso-caloric, but with different intervals of sitting and executing moderate physical activity by treadmill walking corresponding to 60-65% of their individual VO2max values, estimated from the individual's pre-test. The volume of sedentary- and physical activity time will be identical in each trial condition. Blood samples will be taken and blood pressure measured every 30 minutes. The visits for main testing will be separated by a washout period of minimum 5 days, and women will be tested in the follicular phase.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control condition (Experimental): Control condition: Sitting from 8 am until 3pm.
  Interventions: Behavioral: Sedentary breaks
- Condition 1 (Experimental): Condition 1: 35 minutes of treadmill walking followed by sitting until hour 7 is reached
  Interventions: Behavioral: Sedentary breaks
- Condition 2 (Experimental): Condition 2: 2.5 minutes of treadmill walking for every 30 minutes until hour 7 is reached.
  Interventions: Behavioral: Sedentary breaks
- Condition 3 (Experimental): Condition 3: 5 minutes of treadmill walking every 60 minutes, until hour 7 is reached.
  Interventions: Behavioral: Sedentary breaks

INTERVENTIONS:
Behavioral: Sedentary breaks — Interrupting sitting with different frequencies of walking/jogging at moderate intensity.

SUMMARY:
The knowledge gap on sedentary behavior and sedentary breaks includes whether detrimental effects of sedentary behavior can be fully attenuated by 1.) sedentary breaks 2.) physical activity or 3.) both combined. Specifically, when breaking sedentary time which physical activity pattern- and intensity modifies the negative effects of sedentary behavior on glucose- and lipid metabolism? This lack of quantitative evidence calls for prospective experimental studies investigating the physiological and biological impacts of sedentary behavior, as well as the effectiveness of different strategies to reduce sedentary time. Thus, quantifying effects of the intensity, frequency, volume and investigating the patterns of sedentary breaks and/or physical activity on predefined outcomes is of importance.

Aims:

Our primary aims are to investigate the effects of breaking up sedentary time on glucose- and lipid metabolism and thus examine whether pattern for sedentary bouts and breaks and physical activity intensity during sedentary breaks matter. Specifically, the aims of the PhD-project are to provide knowledge on the following questions:

• How does different patterns of accumulation of sedentary bouts and breaks acutely influence glucose- and lipid metabolism under iso-caloric conditions?

DETAILED DESCRIPTION:
The participants will undergo 4 different trial conditions of which all are iso-caloric, but with different intervals of sitting and executing moderate physical activity by treadmill walking corresponding to 45-55% of their individual VO2max/peak values, estimated from the individual's pre-test. The total duration of sedentary- and physical activity time will be identical in each trial condition. This study has a is randomized cross-over design. If found eligible from step 1 and 2 in the inclusion process, participants will be invited to a final screening day in our lab. Eligible participants then consenting to joining the study will continue on to 4 trial days. Due to possible acute rise in insulin for up to 48 hours, a 5-14 day washout period between trials will be used to avoid carryover effects. In the washout periods between experimental conditions the participants will resume their habitual life activities and behaviours, i.e., diet and physical activity patterns. However, from visit 2, during washout the participants will wear accelerometers (ActiGraph GTX3+, Pensacola, FL) during waking hours to objectively measure sedentary time and physical activity. Average sedentary time (hour/day) and time spent in , light-, moderate- and vigorous physical activity intensity (min/day) will be derived. During the main trial days, the participants may read or work on a personal computer during the sedentary time in the respective trial conditions. The sample size calculations with glucose as the primary outcome, are based on the study by Dunstan et al. (2012). They estimated that 19 paired observations were needed to secure a power of 0.90 in order to detect the smallest expected effect size between the interventions, when using a two-tailed test with a significance level of 5%. To account for the possibility of dropouts the sample size in the present project is set to recruit 30 participants, with 25 participants completing the trials, and thus planning for 80% power

ELIGIBILITY:
Inclusion Criteria:

* Predominantly sedentary occupation.
* Physical activity: equal or less tham 150 minutes /week
* Nonobese. Central adiposity: Waist circumference equal or less than 102 cm for men and equal or less than < 88 cm for women. BMI < 30 km·m2

Exclusion Criteria:

* Shift-work
* Smoking
* Pregnancy
* Current use of medication, except from hormonal contraceptives.
* No presence of any co-morbidity (e.g. diabetes type 2, cardiovascular or cardiorespiratory disease, or other conditions known to affect carbohydrate and lipid metabolism - thyroid-, -liver or kidney).
* Systolic /diastolic resting blood pressure: > 140/90 mmHg
* Fasting blood glucose concentration: > 6.1 mmol/L
* Abnormal total cholesterol, LDL, LDL or triglyceride concentrations (> 50% above recommendations)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incremental areas under the curve (iAUC) for glucose | The iAUC for glucose will be assessed during the procedure and consist of measures every 30 minute throughout the trial (420 minutes)
  During each of the trial conditions blood samples will be taken in the fasted state in the morning and then every 30 minutes of the trials (total 420minutes) through a peripheral venous catheter. We will then calculate the iAUC for glucose for each of the trial condition and compare the different trial conditions with the control condition

SECONDARY OUTCOMES:
iAUC analyses for insulin, c-peptide, triglycerides and lipids | The iAUC for the secondary outcomes will be assessed during the procedure and consist of measures every 30 minute throughout the trial (420 minutes)
  During each of the trial conditions blood samples will be taken in the fasted state in the morning and then every 30 minutes of the trials (total 420minutes) through a peripheral venous catheter. We will then calculate the iAUC for glucose for each of the trial condition and compare the different trial conditions with the control condition
Cognitive function - Trail making test A and B | The cognitive measures will be performed during the procedure (at approx 400 minutes)
  Cognitive function tasks will be performed, and cognitive function will be assessed by Trail making test A and B,
Cognitive function - Stroop-test. | The cognitive measures will be performed during the procedure (at approx 400 minutes)
  Cognitive function tasks will be performed, and cognitive function will be assessed by T Stroop-test.

CONTACTS AND LOCATIONS:
Overall Officials: Jostein Steene-Johannessen, Professor, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sports Sciences, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No